CLINICAL TRIAL: NCT03936140
Title: The Effect of Iloprost on Arterial Oxygenation and Shunt Fraction During One-lung Ventilation for Lung Surgery
Brief Title: The Effect of Iloprost on Oxygenation During One-lung Ventilation for Lung Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Wonjung Hwang, Assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC14MISI0880
Record Dates: First submitted 2019-04-08; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Iloprost 10 (Experimental): Iloprost 10μg of inhaled iloprost (Ventavis®)
  Study drug was inhaled to ventilated lung through a nebulized system in inspiratory limb after one-lung ventilation in the lateral decubitus position.
  Interventions: Drug: Inhaled iloprost
- Iloprost 20 (Experimental): Iloprost 20μg of inhaled iloprost (Ventavis®)
  Study drug was inhaled to ventilated lung through a nebulized system in inspiratory limb after one-lung ventilation in the lateral decubitus position.
  Interventions: Drug: Inhaled iloprost
- Distilled water (Placebo Comparator): Distilled water
  Study drug was inhaled to ventilated lung through a nebulized system in inspiratory limb after one-lung ventilation in the lateral decubitus position.
  Interventions: Drug: Distilled water

INTERVENTIONS:
Drug: Inhaled iloprost — Study drug was inhaled to ventilated lung through a nebulized system in inspiratory limb after one-lung ventilation in the lateral decubitus position.
  Arms: Iloprost 10; Iloprost 20
Drug: Distilled water — Study drug was inhaled to ventilated lung through a nebulized system in inspiratory limb after one-lung ventilation in the lateral decubitus position.
  Arms: Distilled water

SUMMARY:
During one-lung ventilation in patients undergoing thoracic surgery, the persistent flow in the non-ventilated lung increases intrapulmonary shunt and decreases systemic arterial oxygenation. This prospective, randomized, double blind study was conducted to evaluate the effects of inhaled iloprost during one-lung ventilation on arterial oxygenation and shunt fraction during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective video-assisted thoracoscopic surgery (VATS) lobectomy
* 20 < age < 75
* American Society of Anesthesiologists (ASA) classification I~III

Exclusion Criteria:

* ASA classification IV
* New York Heart Association (NYHA) class III~IV
* Severe obstructive lung disease / restrictive lung disease
* Pulmonary hypertension
* End-stage organ disease (i.e. hepatic failure, renal failure)
* Arrhythmia
* Previous history of thoracic surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
PaO2(partial pressure of arterial oxygen) | 30 min after treatment
  ABGA
Pulmonary shunt fraction | 30 min after treatment
  Qs/Qt = (CcO2-CaO2) / (CcO2-CvO2)

CONTACTS AND LOCATIONS:
Overall Officials: Wonjung Hwang, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided